CLINICAL TRIAL: NCT06707376
Title: Early Kangaroo Mother Care Versus Standard Neonatal Nursing Practices: A Randomized Controlled Trial on Survival and Nursing Outcomes in Preterm Infants (<2000 g) With Mild to Moderate Respiratory Distress
Brief Title: Early Kangaroo Care vs. Standard Neonatal Practices: Impact on Survival and Outcomes in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Nadia Elsharkawy, Associtae Professor, Jouf University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 547-10-2024
Record Dates: First submitted 2024-11-20; First posted 2024-11-27 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Kangaroo-Mother Care; Preterm Infants
Keywords: Kangaroo-Mother Care; Neonatal Nursing Practices; Preterm Infants

STUDY DESIGN:
Intervention Model Description: Early Kangaroo Mother Care Group:
  * Initiation of KMC within 24 hours of birth.
  * Continuous skin-to-skin contact for at least 8 hours per day, with gradual increase based on infant tolerance.
  * Support for exclusive breastfeeding or expressed breast milk feeding.
  * Ongoing assessment and support from trained neonatal nurses and lactation consultants.
  Control Group:
  * Standard neonatal nursing practices, including incubator care, intermittent holding, and feeding as per clinical guidelines.
  * Respiratory support as needed based on the severity of respiratory distress.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomly assigned to either the Early Kangaroo Mother Care group or control group using a computer-generated randomization sequence with block sizes of varying lengths to ensure allocation concealment and they are unaware of which group they have been assigned to as well as the outcome assessor is unaware
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Kangaroo Mother Care Group (Experimental): Early Kangaroo Mother Care Group:
  * Initiation of KMC within 24 hours of birth.
  * Continuous skin-to-skin contact for at least 8 hours per day, with gradual increase based on infant tolerance.
  * Support for exclusive breastfeeding or expressed breast milk feeding.
  * Ongoing assessment and support from trained neonatal nurses and lactation consultants.
  Interventions: Other: Early Kangaroo Mother Care
- Control Group (No Intervention): Control Group:
  * Standard neonatal nursing practices, including incubator care, intermittent holding, and feeding as per clinical guidelines.
  * Respiratory support as needed based on the severity of respiratory distress.

INTERVENTIONS:
Other: Early Kangaroo Mother Care — * Initiation of KMC within 24 hours of birth.
  * Continuous skin-to-skin contact for at least 8 hours per day, with gradual increase based on infant tolerance.
  * Support for exclusive breastfeeding or expressed breast milk feeding.
  * Ongoing assessment and support from trained neonatal nurses and lactation consultants.
  Arms: Early Kangaroo Mother Care Group

SUMMARY:
This study aims to evaluate the efficacy of Early Kangaroo Mother Care (KMC) compared to standard neonatal nursing practices in improving survival rates and nursing outcomes among preterm infants weighing less than 2000 grams with mild to moderate respiratory distress. Utilizing a randomized controlled trial design, the research will be conducted in neonatal intensive care units (NICUs) across selected hospitals. Primary outcomes include infant survival rates, incidence of complications, and measures of maternal-infant bonding. Secondary outcomes involve nursing practices, caregiver satisfaction, and long-term developmental milestones. The use of validated, free assessment tools will ensure reliability and accessibility. Findings from this study are expected to inform best practices in neonatal care, potentially leading to improved health outcomes for preterm infants.

DETAILED DESCRIPTION:
Preterm birth, defined as delivery before 37 weeks of gestation, is a leading cause of neonatal morbidity and mortality worldwide. Infants weighing less than 2000 grams are particularly vulnerable to complications, including respiratory distress syndrome (RDS), which can significantly impact survival rates and long-term development. Traditional neonatal nursing practices focus on providing respiratory support, maintaining body temperature, and ensuring adequate nutrition. However, emerging evidence suggests that Kangaroo Mother Care (KMC), which emphasizes skin-to-skin contact and exclusive breastfeeding, may offer superior outcomes for preterm infants.

Kangaroo Mother Care (KMC) KMC involves continuous skin-to-skin contact between the mother and infant, promoting thermal regulation, enhancing breastfeeding, and fostering maternal-infant bonding. Studies have indicated that KMC can reduce mortality rates, lower the incidence of infections, and improve neurodevelopmental outcomes. Despite its benefits, the implementation of KMC varies across healthcare settings, and its comparative effectiveness against standard neonatal care practices warrants further investigation.

Objectives

* To compare the survival rates of preterm infants (<2000 g) with mild to moderate respiratory distress receiving early KMC versus standard neonatal nursing practices.
* To evaluate the impact of early KMC on nursing outcomes, including maternal-infant bonding and breastfeeding rates.
* To assess the feasibility and acceptability of implementing early KMC in NICUs.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born at <37 weeks of gestation.
* Birth weight <2000 grams.
* Diagnosed with mild to moderate respiratory distress (based on clinical criteria such as respiratory rate, oxygen saturation levels, and need for respiratory support).

Exclusion Criteria:

* Infants with severe respiratory distress requiring mechanical ventilation.
* Infants with congenital anomalies or other significant health issues.
* Mothers unable or unwilling to provide KMC (e.g., due to medical conditions, lack of willingness).

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Survival Rates | Up to 24 weeks
  Survival Rates will be the proportion of preterm infants who survive following the implementation of KMC, a practice emphasizing continuous skin-to-skin contact and exclusive breastfeeding.
  For infants weighing less than 2000 grams, KMC has been associated with reduced mortality, particularly in low-resource settings where conventional neonatal care may be limited. By promoting physiological stability, enhancing maternal bonding, and reducing the risk of severe complications like infections and hypothermia, KMC offers a cost-effective and impactful approach to improving survival outcomes in this vulnerable population.
Incidence of Complications | Up to 24 weeks
  Incidence of Complications Including infections, intraventricular hemorrhage, and necrotizing enterocolitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital T, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Derived] Ramadan OME, Alshammari AM, Alruwaili AN, Elsharkawy NB, Alhaiti A, Baraka NIM. Transforming neonatal nursing: a randomized controlled trial comparing kangaroo care and standard protocols for survival in preterm infants with respiratory distress syndrome. BMC Nurs. 2025 Apr 16;24(1):430. doi: 10.1186/s12912-025-03088-8. PMID 40241073